CLINICAL TRIAL: NCT05123989
Title: Evaluating the Impact of Personalized Move Goals in a Mobile App on Physical Activity
Brief Title: Evaluating the Impact of Personalized Move Goals on Physical Activity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Welltory Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: WELLTORY-CT001
Record Dates: First submitted 2021-10-25; First posted 2021-11-17 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-05

CONDITIONS: Sedentary Lifestyle; Physical Activity
MeSH Terms: conditions — Sedentary Behavior; Motor Activity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Personalized move goals (Experimental): Participants will be sent daily messages in the Welltory mobile app with personalized move goals that are based on each participant's historical physical activity data and their daily wellbeing
  Interventions: Behavioral: Personalized move goals
- Constant move goals (Active Comparator): Participants will be sent daily messages in the Welltory mobile app with a static move goal of 10,000 steps per day
  Interventions: Behavioral: Constant move goals
- No intervention (No Intervention): Participants will not be sent any messages with move goals in the Welltory mobile app

INTERVENTIONS:
Behavioral: Personalized move goals — Personalized move goals delivered by the Welltory mobile app
  Arms: Personalized move goals
Behavioral: Constant move goals — Static move goal delivered by the Welltory mobile app
  Arms: Constant move goals

SUMMARY:
The purpose of this study is to evaluate the impact of personalized move goals in the Welltory mobile app on daily step count among adults from 30 to 65 years old. The study also aims to assess how personalized move goals impact workout quality and frequency.

DETAILED DESCRIPTION:
The Welltory app sends users messages with move goals to help people move smarter. Adapted daily based on each user's historical data and overall wellbeing, Welltory's move goals gradually increase physical activity levels, motivating sedentary people to move more without demanding drastic lifestyle changes.

This randomized controlled study will assess if messages with personalized move goals in the Welltory mobile app help increase physical activity among adults.

Participants include individuals aged 30-65 who use iPhones, wear an Apple Watch, and lead sedentary lifestyles (their median daily step count does not exceed 6,000). Participants are selected among active Wellotry mobile app users who had previously not received any messages with move goals.

All participants are randomly assigned to 3 groups:

* Participants in group 1 receive daily messages with personalized move goals in the Welltory mobile app. Personalized move goals are computed based on each participant's historical physical activity data and their daily wellbeing.
* Participants in group 2 receive daily messages with a static move goal of 10,000 steps per day in the Welltory mobile app.
* Participants in group 3 use the Welltory mobile app but don't receive any messages with move goals.

For all participants, steps and workouts are automatically registered by their Apple Watch wearable devices and the Welltory mobile app. Additionally, participants regularly measure their body weight and manually record it in the Welltory mobile app.

This study's duration spans a total of 24 weeks for each participant.

ELIGIBILITY:
Inclusion Criteria:

* Using an iPhone smartphone
* Using an Apple Watch
* Willing to use the Welltory app every day for 6 months
* Median daily step count is less than 6,000 in the month before the beginning of this study

Exclusion Criteria:

* Already participating in another physical activity study
* Known medical conditions or physical problems that require special attention in an exercise program
* Pregnant/gave birth in the past 6 month

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-02-01 (Estimated); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Average Steps per Day at 4 weeks | Baseline, 4 weeks
Change from Baseline Average Steps per Day at 8 weeks | Baseline, 8 weeks
Change from Baseline Average Steps per Day at 12 weeks | Baseline, 12 weeks
Change from Baseline Average Steps per Day at 24 weeks | Baseline, 24 weeks

SECONDARY OUTCOMES:
Change from Baseline Body Weight at 12 weeks | Baseline, 12 weeks
  Body weight in kilograms
Change from Baseline Body Weight at 24 weeks | Baseline, 24 weeks
  Body weight in kilograms
Workouts at 4 weeks | 4 weeks
  Total number of workouts over 20 minutes during first 4 weeks of intervention
Workouts at 8 weeks | 8 weeks
  Total number of workouts over 20 minutes during first 8 weeks of intervention
Workouts at 12 weeks | 12 weeks
  Total number of workouts over 20 minutes during first 12 weeks of intervention
Workouts at 24 weeks | 24 weeks
  Total number of workouts over 20 minutes during 24 weeks of intervention
Active calories during workouts at 4 weeks | 4 weeks
  All active calories burned during workouts over 20 minutes
Active calories during workouts at 8 weeks | 8 weeks
  All active calories burned during workouts over 20 minutes
Active calories during workouts at 12 weeks | 12 weeks
  All active calories burned during workouts over 20 minutes
Active calories during workouts at 24 weeks | 24 weeks
  All active calories burned during workouts over 20 minutes

IPD SHARING:
Plan to Share IPD: No